CLINICAL TRIAL: NCT01846663
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial To Evaluate The Efficacy, Safety, And Pharmacokinetics Of Rifaximin 550 Mg In Subjects With Severe Hepatic Impairment And Overt Hepatic Encephalopathy
Brief Title: Efficacy, Safety, And Pharmacokinetics Of Rifaximin In Subjects With Severe Hepatic Impairment And Hepatic Encephalopathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was determined to be infeasible.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RFHE4043
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy; Liver Failure; Hepatic Insufficiency; Liver Diseases; Brain Diseases; Rifaximin; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Failure; Hepatic Insufficiency; Liver Diseases; Brain Diseases; Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifaximin (Experimental): Rifaximin, oral, 550 mg BID, 6 months of treatment
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Placebo, oral, 0 mg BID, 6 months of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo, oral, 0 mg BID, 6 months of treatment
  Arms: Placebo
Drug: Rifaximin — Rifaximin, oral, 550 mg BID, 6 months treatment
  Other Names: XIFAXAN® Tablets
  Arms: Rifaximin

SUMMARY:
The purpose of the study is to evaluate the safety of Rifaximin or placebo in subjects with severe hepatic impairment and Hepatic Encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breast feeding female ≥ 18 years old
* In remission from demonstrated overt HE
* Had ≥1 episode of overt HE associated with liver disease within the last 6 months
* MELD score of ≥ 19
* Has a close family member or other personal contact who is familiar with the subject's HE, can provide continuing oversight to the subject and is willing to be available to the subject during the conduct of the trial

Exclusion Criteria:

* HIV
* History of tuberculosis infection
* Chronic respiratory insufficiency
* Current infection and receiving antibiotics
* Renal insufficiency requiring dialysis
* Active spontaneous bacterial peritonitis infection
* Intestinal obstruction or has inflammatory bowel disease
* Active malignancy within the last 5 years
* Current GI bleeding or has had a GI hemorrhage within past 3 months
* Anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04-03 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Ph.D., Study Director — Bausch Health Americas, Inc.
Locations (28):
- United States (28):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Research, Phoenix, Arizona
  - University Of Arizona Liver Research Institute, Tucson, Arizona
  - Southern California Liver Centers, Coronado, California
  - UCSD Clinical & Translational Research Institute, La Jolla, California
  - Loma Linda University Medical Center Transplantation Institute, Loma Linda, California
  - University of Southern Califorina Keck School Of Medicine, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of Colorado Denver, Aurora, Colorado
  - Salix Site, New Haven, Connecticut
  - Salix Site, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northwestern University-Comprehensive Transplant Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Tulane Abdominal Transplant Research Office, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Salix Site, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Brook Army Medical Center, Fort Sam Houston, Texas
  - Salix Site, Galveston, Texas
  - The Methodist Hospital, Houston, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - VCU/MCV Health Systems, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifaximin | Placebo
Started | 3 | 3
Completed | 0 | 1
Not Completed | 3 | 2
Not completed — Hepatic encephalopathy breakthrough | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Hepatic Encephalopathy (HE) Breakthrough Episode
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

2. Secondary Outcome: Proportion of Participants With HE-related Hospitalization
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Rifaximin | Placebo
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=3) | Placebo (N=3)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0
Septic shock (Infections and infestations) | 1 (1) | 0
Sepsis (Infections and infestations) | 1 (1) | 0
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1 (1)
Urinary tract infection (Infections and infestations) | 0 | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=3) | Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0
Ammonia increased (Investigations) | 1 (1) | 0
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0
Anosmia (Nervous system disorders) | 0 | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 | 1
Dysesthesia (Nervous system disorders) | 0 | 1 (2)
Dysgeusia (Nervous system disorders) | 0 | 1 (1)
Dyslipidemia (Metabolism and nutrition disorders) | 1 (1) | 0
Escherichia infection (Infections and infestations) | 0 | 1 (1)
Fatigue (General disorders) | 1 (1) | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypothermia (General disorders) | 1 (1) | 0
Insomnia (Psychiatric disorders) | 0 | 1
International normalized ratio increased (Investigations) | 0 | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Edema peripheral (General disorders) | 1 (1) | 0
Prothrombin time prolonged (Investigations) | 0 | 1 (1)
Tremor (Nervous system disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.